CLINICAL TRIAL: NCT01840995
Title: The Effect of Stellate Ganglion Block on Intracranial Pressure Predicted by Ultrasonographic Assessment of Optic Nerve Sheath Diameter
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2013-0078
Record Dates: First submitted 2013-04-19; First posted 2013-04-26 (Estimated); Last update posted 2015-01-28 (Estimated); Status verified 2015-01

CONDITIONS: Pain; Intracranial Pressure
Keywords: stellate ganglion block
MeSH Terms: conditions — Pain

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- stellate ganglion block: Patients receiving stellate ganglion block at our pain management clinic
  Interventions: Procedure: ultrasonographic measurement of optic nerve sheath diameter

INTERVENTIONS:
Procedure: ultrasonographic measurement of optic nerve sheath diameter — A thick layer of gel is applied on the upper closed eyelid. The linear 13- to 6-MHz ultrasound probe is then placed in the gel, without exerting pressure on the eye. Two measurements are taken for each optic nerve: one in the transverse plane, with the probe being horizontal, and one in the sagittal plane, with the probe being vertical. The final ONSD is the mean of these measurements.

SUMMARY:
The stellate ganglion block increase cerebral blood flow, as the consequence of that, it has the potential to cause an increase of intracranial pressure (ICP). Previous studies have proposed that ultrasonographic measurements of the optic nerve sheath diameter (ONSD) correlate with signs of increased ICP. Therefore, this study is aim to confirm the increased ICP by ultrasonographic measurement of ONSD after the stellate ganglion block.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (20-70 years of age)
* who were scheduled to receive stellate ganglion block at our pain management clinic

Exclusion Criteria:

* Patients with previous history of neurologic disease, carotid disease, transient ischemic attack, ocular disease and ocular surgery
* Patients with coagulation disorder
* Patients with severe obesity
* Patients with severe cardiovascular or pulmonary disease
* Patients with cognitive deficits or psychiatric illness

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were scheduled to receive stellate ganglion block at our pain management clinic
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2013-04; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
ultrasonographic measurement of optic nerve sheath diameter | 15 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, Seoul, South Korea

REFERENCES:
- [Background] Dubost C, Le Gouez A, Jouffroy V, Roger-Christoph S, Benhamou D, Mercier FJ, Geeraerts T. Optic nerve sheath diameter used as ultrasonographic assessment of the incidence of raised intracranial pressure in preeclampsia: a pilot study. Anesthesiology. 2012 May;116(5):1066-71. doi: 10.1097/ALN.0b013e318246ea1a. PMID 22258019